CLINICAL TRIAL: NCT04462432
Title: Spatiotemporal Characteristics and Multi-body Dynamics Modeling of Gait Touch Information After Anterior Cruciate Ligament Rupture and Reconstruction
Brief Title: Spatiotemporal Characteristics and Multi-body Dynamics Modeling Information After ACL Rupture and Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OR003
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; gait analysis; plantar pressure; multi-body dynamics modeling
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior Cruciate Ligament injury and reconstruction group: According to the previous clinical diagnosis, volunteers who has never suffered the Anterior Cruciate Ligament injury.
  Interventions: Other: no intervention
- normal control group: According to the previous clinical diagnosis, volunteers who has never suffered the lower extremity sports injuries.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study, with no intervention.

SUMMARY:
High incidence rate of knee osteoarthritis and gait analysis are important for early assessment of biomechanics. ACL injury is an ideal clinical model for studying knee osteoarthritis.

To clarify the mechanism between the biomechanical status of knee joint and the change of gait touch information, and to provide scientific basis for quantifying and evaluating the biomechanical status of knee joint in dynamic load-bearing state.

DETAILED DESCRIPTION:
Purpose: To clarify the relationship between the normal and abnormal biomechanical status of the knee joint and the gait touch information, and to establish the biomechanical evaluation model of the knee joint during walking or jogging, taking into account the comprehensive effects of sports parameters, individual attribute parameters and other factors. An automatic analysis and expert diagnosis system was established to evaluate the biomechanics of knee joint.

Methods: 50 young male (23-35 years old) healthy volunteers and 100 patients with unilateral simple ACL rupture who need surgical treatment were recruited, 150 subjects in total. Three tests were performed before surgery, at the end of the 24th and 48th weeks after surgery. All were tested with three-dimensional gait analysis, dynamic plantar pressure measurement and isokinetic muscle strength during walking, jogging, emergency stop and take-off, side cut.

Outcome evaluation indicators and statistical methods: Two-way ANOVA method of repeated measurement was used, the left and right sides and different rehabilitation time were used as the variables of repeated measurement: the biomechanics of the lower limb joint and the change of the biological characteristics of the gait touch information were analyzed. Three dimensional gait analysis and computer-aided analysis of gait touch information were used to study the changes of ACL rupture and reconstruction. Based on the information of gait touch, taking into account the comprehensive effects of sports parameters, individual attribute parameters and other factors, a biomechanical evaluation model of knee joint during walking or jogging is established, which provides the exact basis for quantifying the information of gait touch and evaluating the biomechanical state of knee joint after ACL rupture and reconstruction under dynamic load-bearing state, and establishes a clinical practical automatic analysis and expert diagnosis system of gait touch information to evaluate the biomechanics of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital.
* With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures).
* All participants have no known disorders or diseases other than ACL rupture.

Exclusion Criteria:

* Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion criteria: Age: 18-35 years old. Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital. With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures). All participants have no known disorders or diseases other than ACL rupture.
  Exclusion criteria: Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
walking speed | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
walking speed | at 24th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
walking speed | at 48th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
ground reaction force | at 24th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
ground reaction force | at 48th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
knee flexion angle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
knee flexion angle | at 24th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
knee flexion angle | at 48th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | at 24th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | at 48th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee flexion in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee flexion in the gait cycle | at 24th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee flexion in the gait cycle | at 48th weeks after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | On the day of enrollment, at 24th and 48th weeks after Anterior Cruciate Ligament reconstruction.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No